CLINICAL TRIAL: NCT06928025
Title: Effectiveness of Animation-Based Training Given to Elderly Patients Who Will Have Coronary Artery Bypass Graft Surgery on Their Pain, Fear, Anxiety and Self-Care Management: Randomized Control Study
Brief Title: Effectiveness of Animation-Based Education Given to Elderly Patients Undergoing Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşegül Sena Pirgaip Yavuz (Other)
Responsible Party: Sponsor-Investigator, Ayşegül Sena Pirgaip Yavuz, Clinical Nurse, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AYavuz
Record Dates: First submitted 2025-03-30; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Surgery
Keywords: Nursing; elderly patient; anxiety; self-care management; pain; fear; coronary artery bypass surgery
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animation Based Education (Experimental): Experimental: Patients in the experimental group will be given animation-based video training with a laptop one day before the surgery. The animation-based video training lasts 8 minutes and 35 seconds in total.
  Patient Information Form, Self-Care Management in Chronic Diseases Scale, Visual Analog Scale, Hospital Anxiety Depression Scale, Surgical Fear Scale (Turkish Version) will be applied.
  Interventions: Procedure: Preoperative Education
- Control (No Intervention): Control: In the preoperative period, no training will be given by the researcher to the patients constituting the control group. Patients in this group will receive the routine training of the clinic before surgery. Patient Information Form, Self-Care Management in Chronic Diseases Scale, Visual Analog Scale, Hospital Anxiety Depression Scale, Surgical Fear Scale (Turkish Version) will be applied.

INTERVENTIONS:
Procedure: Preoperative Education — animation-based education for elderly patients before coronary artery bypass graft surgery Before coronary artery bypass graft surgery, the scenario prepared based on the literature information including introduction of the service, preparation for surgery, monitoring, drug treatment and applications, deep breathing and cough exercise, spirometer use, operation time, postoperative period and care, patient pain management and intubation process will be given as animation-based video training. The effects of this on postoperative pain, fear, anxiety and self-care management will be evaluated.
  Arms: Animation Based Education

SUMMARY:
It was conducted to measure the effectiveness of animation-based training given to elderly patients who will undergo coronary artery bypass graft surgery on the patients' pain, fear, anxiety and self-care management.

The study will be completed with 72 participants, 35 experimental and 37 control.

As a randomization method, simple randomization method will be used to ensure equal number of samples in the two groups, and patients will be verbally informed about the study and written informed consent will be obtained from the patients who agree.

In this study, the effectiveness of animation-based training given to elderly patients undergoing coronary artery bypass graft surgery on pain, fear, anxiety and self-care management will be evaluated.

DETAILED DESCRIPTION:
Experimental: Patients in the experimental group will be given animation-based video training with a laptop one day before the surgery. The animation-based video training lasts 8 minutes and 35 seconds in total.

Patient Information Form, Self-Care Management in Chronic Diseases Scale, Visual Analog Scale, Hospital Anxiety Depression Scale, Surgical Fear Scale (Turkish Version) will be applied.

Control: In the preoperative period, no training will be given by the researcher to the patients constituting the control group. Patients in this group will receive the routine training of the clinic before surgery. Patient Information Form, Self-Care Management in Chronic Diseases Scale, Visual Analog Scale, Hospital Anxiety Depression Scale, Surgical Fear Scale (Turkish Version) will be applied.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older,
* No diagnosed functional disability,
* First scheduled coronary artery bypass graft surgery,
* Those who volunteered to participate in the study

Exclusion Criteria:

* Urgent cases,
* Cases with additional surgical procedures

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Patient Information Form | Up to 24 weeks
  The personal information form used for data collection consists of demographic characteristics of the individuals such as age, gender, marital status, occupation, educational status, employment status, as well as questions including health-related conditions of the patients such as chronic diseases, whether they have had surgery before or not.

SECONDARY OUTCOMES:
Self-Care Management Scale in Chronic Diseases | Up to 24 weeks
  Self-Care Management-Protection (SCMP-G) After Jones and Preuett defined the concept of self-care management process (SCMP), the validity of SCMP was tested and the characteristics of the protection concept were explained and added.While developing the SCMP-G scale, two types of protection concepts were defined.These concepts were determined as self-protection and social protection and formed two sub-dimensions of the scale. The self-protection sub-dimension consists of items numbered 2, 6, 8, 11, 15, 18, 19, 20, 22, 23 and 25-34, while the social protection sub-dimension consists of items numbered 1, 3-5, 7, 9, 10, 12-14, 16, 17, 21, 24 and 35.The scale has a format that is evaluated between 5 (Strongly Agree) and 1 (Strongly Disagree).The higher the score, the higher the level of self-care management.The Cronbach's Alpha of the self-care management scale in chronic patients is 0.85. The Cronbach's Alpha for this study was 0.89.

OTHER OUTCOMES:
Hospital Anxiety Depression Scale | Up to 24 weeks
  The Hospital Anxiety and Depression Scale is a scale consisting of a total of 14 items. Odd numbered items assess anxiety and even numbered items assess depression. The scale has a four-point Likert-type structure and the score range of the items is between 0 and 3. The total scores of the subscales are calculated by summing the scores of the related items. To calculate the anxiety subscale score, the scores of the 1st, 3rd, 5th, 7th, 7th, 9th, 11th and 13th items should be summed, while the scores of the 2nd, 4th, 6th, 8th, 10th, 12th and 14th items should be summed for the depression subscale score. Individuals who score above these cut-off points should be considered in the risk group. The Cronbach's Alpha of the scale is 0.81. The Cronbach's Alpha of this study was 0.89.
Surgical Fear Scale | Up to 24 weeks
  The surgical fear scale was developed in 2014 to determine the fear levels of patients undergoing elective surgery due to the short- and long-term consequences of the surgical operation.The SCS is an 11-point scale consisting of 8 items and scored from 0 to 10. Each item is scored from 0 (not at all afraid) to 10 (very afraid). The scale has two subdimensions; Surgical Fear Scale Short-Term (SCS-S-S) and Surgical Fear Scale Long-Term (SCS-L). Items 1-4 on the scale show short-term outcomes, while items 5-8 show long-term outcomes. The subscale score is obtained by adding the scores of the four items in the sub-dimensions of the scale, and the total score of the scale is obtained by adding the scores of the two sub-scales.The lowest score in the subscales is 0 and the highest score is 40. Fear of surgery increases in parallel with the score obtained. The Cronbach's Alpha value of the scale is 0.93. The Cronbach's Alpha value of this study was found to be 0.93.
Visual Analog Scale | Up to 24 weeks
  It is a table used to assess pain. The Visual Analog Scale, developed by Cline and colleagues, is a 10 cm long, horizontal or vertical ruler that allows the assessment of pain level on a scale from "no pain" to "unbearable pain". The patient marks their pain on this scale and indicates their pain score.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk Universty, Erzurum, Palandöken, Turkey (Türkiye)